CLINICAL TRIAL: NCT05801042
Title: Comparing the Efficacy of Micro-encapsulated Lactocaseibacillus Rhamnosus Vs Free Probiotic in Powder to Affect Brain Connectivity
Brief Title: Effect of Encapsulated Vs Free Probiotic on Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Brummer (Other)
Responsible Party: Sponsor-Investigator, Robert Brummer, Principal Investigator, Örebro University, Sweden
Organization: Örebro University, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AnaBio
Record Dates: First submitted 2023-02-10; First posted 2023-04-06 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Aging
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Encapsulated probiotic (Experimental)
  Interventions: Dietary Supplement: Encapsulated Lactocaseibacillus rhamnosus
- Non-encapsulated probiotic (Active Comparator)
  Interventions: Dietary Supplement: Non-encapsulated Lactocaseibacillus rhamnosus
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Maltodextrin — Placebo product
  Arms: Placebo
Dietary Supplement: Encapsulated Lactocaseibacillus rhamnosus — Probiotic product
  Arms: Encapsulated probiotic
Dietary Supplement: Non-encapsulated Lactocaseibacillus rhamnosus — Probiotic product
  Arms: Non-encapsulated probiotic

SUMMARY:
Aging is associated with changes in a wide variety of brain networks, including the default mode, saliency attention, and visual networks. Furthermore, current research suggests that a relationship exists between functional connectivity at rest and cognition. Lactocaseibacillus rhamnosus is an ideal strain for the intervention, as it has been show to affect the gut-brain axis, brain function, and behavior. Therefore, the investigators plan to assess resting state functional magnetic resonance imaging (fMRI) to compare changes in brain connectivity between the groups receiving the encapsulate and non-encapsulated Lactocaseibacillus rhamnosus supplements.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedure
2. Age 60-80 years-old
3. Normal weight at the screening defined as BMI range 18.5-31.9
4. Willing to abstain from regular consumption of probiotic supplements or food products containing probiotic bacteria (including fermented food and beverages)
5. Willing to abstain from regular consumption of supplements and medications known to alter gastrointestinal function or inflammatory status during the study

Exclusion Criteria:

1. Diagnosis of type 1 and/or type 2 diabetes
2. Current (or within the last 4 weeks prior to study start) use of probiotic supplementation
3. Immobile (defined as the inability to participate in all study-related procedures)
4. History of complicated gastrointestinal surgery
5. Diagnosed inflammatory bowel disease (IBD)
6. Current diagnosis of psychiatric disease/s or syndromes
7. Current diagnosis of neurodegenerative disease
8. Systemic use of antibiotics and/or steroid medication in the last 4 months prior to inclusion
9. Use of any non-steroidal anti-inflammatory drug (NSAID) more than 3 times a week for the last 2 months
10. Consumption of any NSAID within 7 days of study start
11. Any condition which could substantially interfere with intestinal barrier function (e.g. gluten sensitivity, lactose intolerance, celiac disease, irritable bowel syndrome (IBS), IBD) or in any other way with the outcome of the study, as decided by the principle investigator's discretion
12. Regular smoking, use of snuff, nicotine, cannabidiol narcotics/supplements, or e-cigarette use
13. Drinking more than 9 standard cups of alcohol per week and/or more than 3 standard cups of alcohol per occasion
14. Regular use, for more than three times a week for the last 2 months and/or 7 days prior to inclusion, of medications which according to the principal investigator can have an anti-inflammatory effect or affect in any way the intestinal barrier function or have an impact on the study analysis (such as laxatives, anti-diarrheal, anti-cholinergic, etc.)
15. After being included in the study, starting any medication or treatment that could potentially influence the study participation and/or study analysis
16. Cerebral bleeding or history of cerebral bleeding
17. Claustrophobia
18. In operated apparatus (e.g., pacemaker), as it interferes with MR imaging
19. Aneurysm clips in the head
20. Shunts in the head
21. Grenade-splinter or metal-splinter in the body (e.g., eyes)
22. Metal or electrodes in the body (e.g., temp-catheter, aorta stent, cochlear implant)
23. Comprehensive tooth-implants or prosthesis
24. Operated in the head
25. Operated in the heart
26. Swallowed a video-capsule, which may still be in the GI tract
27. Left-handed

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Brain functional connectivity as measured by resting-state functional magnetic resonance imaging (fMRI) | 6 weeks
  corrected for baseline

SECONDARY OUTCOMES:
Levels of inhibitory neurotransmitter gamma-aminobutyric acid (GABA) in the brain using MR spectroscopy (MRS) | 6 weeks
  corrected for baseline
Cognitive function assessment using the trail making test (TMT) | 6 weeks
  corrected for baseline, scale 0-400 seconds and number of errors, higher scores indicate worse cognition
Cognitive function assessment using digit symbol substitution test (TMT) | 6 weeks
  corrected for baseline, scale 0-93 points, higher scores indicate better cognition
Cognitive function assessment using letter digit substitution test | 6 weeks
  corrected for baseline, scale 0-135 points, higher scores indicate better cognition
Cognitive function assessment using letter comparison test | 6 weeks
  corrected for baseline, scale 0-42 points, higher scores indicate better cognition
Cognitive function assessment using Rey-Auditory Verbal Learning Test | 6 weeks
  corrected for baseline, scale 0-120 points, higher scores indicate better cognition
Cognitive function assessment using N-back task | 6 weeks
  corrected for baseline, higher scores indicate better cognition
Cognitive function assessment using Face-Name Paired Associate Task (FNPA) | 6 weeks
  corrected for baseline, higher scores indicate better cognition
Levels of inflammatory markers (e.g. high sensitivity C-reactive protein (hsCRP), interleukin (IL)-6, tumor necrosis factor (TNF)-alpha) | 6 weeks
  corrected for baseline, unit of measurement concentration given as mg/ml
Levels of inflammatory markers (e.g. high sensitivity C-reactive protein (hsCRP), interleukin (IL)-6, tumor necrosis factor (TNF)-alpha) | 3 weeks
  corrected for baseline, unit of measurement concentration given as mg/ml
Levels of metabolic blood markers (blood fats) | 6 weeks
  corrected for baseline, unit of measurement concentration given as mg/ml
Levels of metabolic blood markers (blood fats) | 3 weeks
  corrected for baseline, unit of measurement concentration given as mg/ml
Levels of neural blood markers (brain derived neurotrophic factor (BDNF), serotonin) | 6 weeks
  corrected for baseline, unit of measurement concentration given as mg/ml
Levels of neural blood markers (brain derived neurotrophic factor (BDNF), serotonin) | 3 weeks
  corrected for baseline, unit of measurement concentration given as mg/ml
Characterisation of lymphocyte subpopulations using flow cytometry | 6 weeks
  corrected for baseline
Faecal samples for evaluation of gut microbiota composition via next-generation sequencing (NGS) | 6 weeks
  corrected for baseline

OTHER OUTCOMES:
Brain stem functional connectivity as measured by resting-state functional magnetic resonance imaging (fMRI) | 6 weeks
  corrected for baseline
Brain structure measured by magnetic resonance imaging (fMRI) | 6 weeks
  corrected for baseline
Characterisation of probiotic bacteria in faecal samples using flow cytometry | 6 weeks
  corrected for baseline
Assessment of psychological health using Hospital Anxiety and Depression Scale (HADS) | 3 weeks
  corrected for baseline, scale 0-42, higher score indicates worse anxiety and depression symptoms
Assessment of psychological health using Hospital Anxiety and Depression Scale (HADS) | 6 weeks
  corrected for baseline, scale 0-42, higher score indicates worse anxiety and depression symptoms
Assessment of psychological health using Pittsburgh Sleep Quality Index (PSQI) | 3 weeks
  corrected for baseline, scale 0-21, higher score indicates worse sleep
Assessment of psychological health using Pittsburgh Sleep Quality Index (PSQI) | 6 weeks
  corrected for baseline, scale 0-21, higher score indicates worse sleep
Assessment of psychological health using Perceived Stress Scale (PSS) | 3 weeks
  corrected for baseline, scale 0-40, higher score indicates more perceived stress
Assessment of psychological health using Perceived Stress Scale (PSS) | 6 weeks
  corrected for baseline, scale 0-40, higher score indicates more perceived stress
Assessment of gastrointestinal health using Gastrointestinal Symptoms Rating Scale (GSRS) | 3 weeks
  corrected for baseline, scale 15-105, higher score indicates more gastrointestinal symptoms
Assessment of gastrointestinal health using Gastrointestinal Symptoms Rating Scale (GSRS) | 6 weeks
  corrected for baseline, scale 15-105, higher score indicates more gastrointestinal symptoms
Cognitive function assessment using the Montreal Cognitive Assessment (MoCA) | 6 weeks
  corrected for baseline, scale 0-30 points, higher scores indicate better cognition
Brain functional connectivity as measured by resting-state functional magnetic resonance imaging (fMRI) | 10-12 weeks
  corrected for baseline
Assessment of psychological health using Hospital Anxiety and Depression Scale (HADS) | 10-12 weeks
  corrected for baseline, scale 0-42, higher score indicates worse anxiety and depression symptoms
Assessment of psychological health using Pittsburgh Sleep Quality Index (PSQI) | 10-12 weeks
  corrected for baseline, scale 0-21, higher score indicates worse sleep
Assessment of psychological health using Perceived Stress Scale (PSS) | 10-12 weeks
  corrected for baseline, scale 0-40, higher score indicates more perceived stress
Assessment of gastrointestinal health using Gastrointestinal Symptoms Rating Scale (GSRS) | 10-12 weeks
  corrected for baseline, scale 15-105, higher score indicates more gastrointestinal symptoms
Brain structure measured by magnetic resonance imaging (fMRI) | 10-12 weeks
  corrected for baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert JM Brummer, MD PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rode J, Hutchinson AN, Chatzopoulou MS, Bleiel SB, Gebresenbet RF, Andersson L, Persson J, Daillere R, Beitz B, Ben Abdallah B, Tingo L, Bergh C, Brummer RJ. Micro-encapsulation differentially impacts probiotic effects on brain structure and function in an elderly population - A randomised placebo-controlled trial. Brain Behav Immun. 2025 Nov;130:106113. doi: 10.1016/j.bbi.2025.106113. Epub 2025 Sep 19. PMID 40976401